CLINICAL TRIAL: NCT06821776
Title: N-of-1 Trial Comparing Prolonged Gastric Feeding to Transpyloric Feeding in Infants with Severe Bronchopulmonary Dysplasia
Brief Title: Gastric Feeding Versus Transpyloric Feeding in Infants with Severe Bronchopulmonary Dysplasia, a Crossover Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-10394-FB
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Bronchopulmonary Dysplasia; Feeding Intolerance
Keywords: BPD
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastric feeding (Active Comparator): Subject will receive 2 weeks of continuous gastric feeding via a feeding tube in the stomach.
  Interventions: Procedure: Gastric feeding
- Transpyloric feeding (Active Comparator): Subject will receive 2 weeks of continuous transypyloric feeding via a feeding tube that passes through the stomach into the first portion of the small intestine.
  Interventions: Procedure: Transpyloric feeding

INTERVENTIONS:
Procedure: Gastric feeding — Subjects will be fed through a feeding tube that empties into the stomach.
  Arms: Gastric feeding
Procedure: Transpyloric feeding — Subjects will be fed through a feeding tube that passes through the stomach and empties directly into the small intestine.
  Arms: Transpyloric feeding

SUMMARY:
Hospitalized infants with severe bronchopulmonary dysplasia (BPD) and feeding intolerance will be randomized to 2 weeks of continuous gastric feeding or continuous transpyoloric feeding. Subjects will crossover after 2 weeks and receive 4 weeks of each feeding mode. Respiratory status will be assessed to determine the optimal feeding mode for each infant.

ELIGIBILITY:
Inclusion Criteria:

* Patients born <32 weeks' gestation
* Currently admitted to the Le Bonheur NICU
* Grad 2 or 3 BPD (positive pressure or intubated at 36 weeks PMA)
* Signs of gastroesophageal reflux, chronic aspiration, or other feeding intolerance.

Exclusion Criteria:

* Known gastrointestinal anomalies
* Unable to tolerate ≥100mL/kg/day enteral feeding
* Congenital anomalies likely to alter feeding techniques
* Surgical feeding tube in place or expected within the next 8 weeks
* Expected to remain hospitalized <8 weeks

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory Severity Score (RSS) | 8 weeks
  RSS (the product of mean airway pressure and oxygen fraction) will be calculated before and after each 2-week intervention block.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weems, MD, Principal Investigator — University of Tennessee
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lillie EO, Patay B, Diamant J, Issell B, Topol EJ, Schork NJ. The n-of-1 clinical trial: the ultimate strategy for individualizing medicine? Per Med. 2011 Mar;8(2):161-173. doi: 10.2217/pme.11.7. PMID 21695041
- [Background] Baker CD, Liptzin DR, Eldredge LC. Transpyloric feeding in severe BPD: a call for prospective trials. J Perinatol. 2024 Jul;44(7):1079. doi: 10.1038/s41372-024-01919-1. Epub 2024 Mar 2. No abstract available. PMID 38431754
- [Background] Levin JC, Kielt MJ, Hayden LP, Conroy S, Truog WE, Guaman MC, Abman SH, Nelin LD, Rosen RL, Leeman KT. Transpyloric feeding is associated with adverse in-hospital outcomes in infants with severe bronchopulmonary dysplasia. J Perinatol. 2024 Feb;44(2):307-313. doi: 10.1038/s41372-024-01867-w. Epub 2024 Jan 13. PMID 38218908
- [Background] Jensen EA, Zhang H, Feng R, Dysart K, Nilan K, Munson DA, Kirpalani H. Individualising care in severe bronchopulmonary dysplasia: a series of N-of-1 trials comparing transpyloric and gastric feeding. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):399-404. doi: 10.1136/archdischild-2019-317148. Epub 2019 Nov 4. PMID 31685527